CLINICAL TRIAL: NCT02808884
Title: Cancer DNA Screening Pilot Study (CANDACE)
Acronym: CANDACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: University of British Columbia (Other); University of Utah (Other); Pathway Genomics (Industry); Boreal Genomics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H16-00519
Record Dates: First submitted 2016-06-07; First posted 2016-06-22 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Intervention Model Description: Blood test screening for all who wish to participant. Additional screening test for those who test positive twice.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Circulating tumor DNA assay- First test - Negative result (Experimental): Once the data is analyzed, participants with a negative result will be sent an email thanking them for their participation and informing them of the negative result.
  Interventions: Genetic: Circulating tumor DNA assay
- Circulating tumor DNA assay - Second test- Negative result (Experimental): Participants whose sample provided a positive result after first test, will be contacted immediately by telephone by an oncologist co-investigator and concurrently sent a letter by mail informing them of the result and asking them to return for a second blood draw. We expect that this communication will happen with about a month of the original blood draw. The letter will include contact information for the study team and the oncologist co-investigators, in case the participant has any questions or concerns at this stage. A requisition form will be sent with the letter. Two 10mL tubes of blood will be drawn at the blood collection visit, to allow repeat testing and confirmation that the mutation is present consistently. Once the data is analyzed, participants with a negative result will be sent an email thanking them for their participation and informing them of the negative result.
  Interventions: Genetic: Circulating tumor DNA assay
- Circulating tumor DNA assay - Second test- Positive result (Experimental): Participants with positive results after first test will be contacted by an oncologist and sent a letter informing them of the result. They will be ask to return for a second blood draw. The letter will include contact info of the study team and the oncologist co-investigators. A requisition form will be sent with the letter. Two 10mL tubes of blood will be drawn to allow repeat testing and confirmation that the mutation is consistently present. Participants whom additional blood sample yields a positive result for the same cancer mutations seen in the first blood draw, will be contacted by an oncologist to explain the results and next steps. This should happen within about a week of the second blood draw. Pending oncological evaluation of the participant and study results, a PET-CT scan with FDG agent, and possibly other tests will be requested. Unless exams suggest otherwise, the default follow-up will be a full body PET-CT.
  Interventions: Genetic: Circulating tumor DNA assay

INTERVENTIONS:
Genetic: Circulating tumor DNA assay — Blood samples will be separated into plasma and cellular fraction including erythrocytes and buffy coat.The plasma fraction will be placed in a separate tube and frozen for subsequent analysis. Frozen plasma samples, de-identified, will be delivered to Pathway Genomics where DNA content will be analyzed with a circulating tumor DNA assay employing the UBC/Boreal Genomics enrichment technology. All of the participants' plasma will be sent to Pathway, where it will be used up in the assay. Circulating tumor DNA assay results (raw sequencing data) from Pathway Genomics will be returned to UBC and analyzed for the presence of cancer mutations. Any samples showing activating mutations above the assay's technical Limit of Detection (LOD) will be called positive. One exception will be made for TP53 mutations that are known to exist in some normal individuals at low levels. For these mutations, a level of 0.1% will be set, above which the sample will be called positive.

SUMMARY:
The investigators have developed an assay that can sensitively and specifically detect DNA mutations circulating in human plasma that may be indicators of the presence of a solid tumor. This study is a pilot study to measure positive and negative predictive values of this assay as an indicator of the presence of a tumor in normal subjects

DETAILED DESCRIPTION:
Participants consenting for the study will be requested to consent for an initial collection of two vials of blood (~ 20 ml total) and to answer questions regarding aspects of their medical history and lifestyle that are relevant to cancer risk. Participants in the study will also be asked to provide consent for follow-up blood samples, and if the confirmatory tests show a positive result, follow-up PET/CT scans and other investigations.

1,000 participants between the ages of 55 and 75 will be enrolled through BC Generations Project. This is a invite-only study.

* Respondents who provide consent and choose to be enrolled in the study will then be directed to an online questionnaire where they will be asked to answer questions regarding their lifestyle and medical history.
* The consent form and questionnaire results will be electronically received at the UBC study site.
* Once participant information has been received at UBC, it will be entered into a password protected spreadsheet on a UBC server. At that point, participants will be sent a requisition form directing them to one of several possible blood collection sites (LifeLabs), where two 10mL blood draws will be collected by a phlebotomist. Blood collections will be paid for by Boreal through a contract with LifeLabs, and will be performed in Streck stabilized cfDNA blood collection tubes (capable of storing blood at room temperature for over a week).
* Once collected, the two blood tubes will be delivered by LifeLabs to BC Cancer Research Center within 24-48 hrs of collection. The tubes will be collected by study staff (within 5 days of the initial blood draw) and transported to UBC, where they will be de-identified and assigned a random identifier (UBC study number). Any personal identification on the tubes will be completely removed, by abrasion if necessary. Identifying information will be entered in a password protected spreadsheet (on a UBC server) linking the participant information to the UBC study number. From this point on, the blood samples, and subsequent fractions and results, will only be identified by the study number. The de-identified tubes will be transported to Boreal Genomics where they will be separated into plasma and cellular fraction including erythrocytes and buffy coat. The non-plasma components of the blood samples will be pooled and subsequently discarded. The plasma fraction will be placed in a separate tube and frozen for subsequent analysis. The original blood tubes (now empty), will be destroyed.
* Frozen plasma samples, now de-identified, will be delivered to Pathway Genomics (San Diego, CA) where DNA content will be analyzed with a circulating tumor DNA assay employing the UBC/Boreal Genomics enrichment technology. All of the participants' plasma will be sent to Pathway, where it will be used up in the assay. Any plasma not consumed in the assay will be destroyed. No plasma, blood or other samples will be stored at either Pathway Genomics or UBC, beyond any temporary storage (1-2 weeks) required to perform the assay.
* Circulating tumor DNA assay results (raw sequencing data) from Pathway Genomics will be returned to UBC and analyzed for the presence of cancer mutations. Any samples showing activating mutations above the assay's technical Limit of Detection (LOD) will be called positive. One exception will be made for TP53 mutations that are known to exist in some normal individuals at low levels. For these mutations, a level of 0.1% will be set, above which the sample will be called positive.
* Once the data is analyzed, participants with a negative result will be sent an email thanking them for their participation and informing them of the negative result.
* Participants whose sample provided a positive result will be contacted immediately by telephone by an oncologist co-investigator and concurrently sent a letter by mail informing them of the result and asking them to return for a second blood draw. The investigators expect that this communication will happen with about a month of the original blood draw. The letter will include contact information for the study team and the oncologist co-investigators, in case the participant has any questions or concerns at this stage. A requisition form will be sent with the letter. Two 10mL tubes of blood will be drawn at the blood collection visit, to allow repeat testing and confirmation that the mutation is present consistently.
* Samples from the additional draw will be treated as described above for the initial samples, with two exceptions. One, the samples will be processed at Boreal Genomics instead of being shipped to Pathway Genomics. Two, some buffy coat DNA (germline DNA) will also be tested for the 96 cancer mutations present on the Boreal panel to detect rare cases where the circulating tumor DNA signal derives from low level germline mutations instead of tumor DNA. This testing will be done at Boreal Genomics and any remaining buffy coat or DNA not consumed in the test will be discarded. Data from the circulating tumor DNA assay and buffy coat test will be returned to UBC and compared to the initial blood result.
* Participants who are found to have a cancer-associated germline mutation during the foregoing testing will be informed by the oncologist co-investigators and will be offered a consultation with the Hereditary Cancer Program at the BC Cancer Agency where they can meet with a medical geneticist for a consultation. If they wish it, these participants would have access to clinically validated retesting for the germline mutation.
* Participants for which the additional blood sample does not yield positive results for cancer mutations, will be contacted by telephone to explain the results.
* Participants for whom the additional blood sample yields a positive result for the same cancer mutations seen in the first blood draw will be contacted by telephone by an oncologist co-investigator, to explain the results and next steps. They will also be sent a letter. The investigators expect this communication to happen within about a week of the second blood draw. Pending oncological evaluation of the participant (see below) and study results, a PET-CT scan with fluorodeoxyglucose (FDG) agent, and possibly other tests will be requested. Unless the oncological exams suggest otherwise, the default follow-up will be a full body PET-CT. The participants undergoing medical imaging scans will be given a requisition form and directed to have the requested scan, which will be paid for by the study sponsor (Boreal Genomics).
* Recognizing that being advised of an abnormal DNA test may cause participants distress, the investigators have committed to (a) complete testing and to contact the participant about the result of 2nd test within 14 days of the blood being drawn; (b) notification of 2nd result (abnormal or normal) being done by phone by the study oncologist (c) pre-booking the follow-up oncological evaluation appointment and offering the participant two options when phoned to advise of the 2nd abnormal result (d) completing the oncological evaluation within 3 weeks of the patient being advised that the 2nd test is abnormal.
* The oncological evaluation will be performed at the Vancouver Centre of the BC Cancer Agency and is likely to include:

  * A full history, including risk factors for cancer and a review of systems to seek symptoms that could be from cancer.
  * A physical examination of:

    - Head and neck, thorax, abdomen, skin, neurological system lymphatic system and rectum. In men: prostate examination. In women: breast and gynecological examinations
  * A whole-body PET-CT scan
  * Standard age-appropriate cancer screening investigations such as the fecal immunochemical test (FIT) for colorectal cancer, Papanicolaou test for cervix cancer and mammography for breast cancer, if they have not been completed, are due, or are overdue.
  * Additional investigations will be guided by the history, physical examination, whole-body PET-CT and standard screening investigations.
  * Investigations may include: complete blood count, liver enzymes, tumour markers, urinalysis, contrast-enhanced MRI, contrast-enhanced CT, as well as endoscopy of the head and neck, bronchi, bladder, upper GI tract and lower GI tract.
* Results of these tests will be returned to the oncologist investigators and to Dr. Marziali and then entered into the study database. The results will be communicated to the participant in writing as well as in person or by phone. The oncologist will refer participants for additional testing and to appropriate clinicians for follow up for additional investigations. The oncologist will also offer a referral of participants to supportive counseling at this stage.
* The results will be communicated to the participant's family physician, if the participant has one, by an oncologist investigator.
* Participants whose investigations detect a potentially malignant mass will have a biopsy, either with imaging guidance, or through referral to an appropriate specialist.
* Participants, whose investigations do not detect a potentially malignant mass, will be informed in writing, as well as in person or by phone that the circulating tumor DNA test gave a false positive result and will be advised to continue with appropriate cancer screening for their age and family history.
* Participants with positive circulating tumor DNA results who are unwilling to undergo further testing including possible PET-CTs will still be offered a follow up visit with the oncologist co-investigator to discuss the results and to offer supportive counseling as described above.
* A year following the initial blood draw, participants will be contacted by email to determine if a cancer diagnosis has been made during that time. For non-responding participants, they will be telephoned and their family physicians will be sent a letter inquiring whether the participant was diagnosed with cancer.

Data collected in this study will be provided to BC Generations Project.

ELIGIBILITY:
Inclusion Criteria:

* Have never been diagnosed with cancer (except for non-melanoma skin cancer)
* Must be able to read and understand a consent form in English
* Be willing to consent to the required blood draws, medical exam and PET-CT scans
* Be willing to consent to any medical data related to this test, the imaging scans, and related follow up, being shared with the study investigators for the following year
* Be in good health and able to donate three tubes of blood
* Must have email
* Must be able to have blood work in the greater Vancouver area

Exclusion Criteria:

* Immunocompromised individuals
* Contra-indications to MRI or PET-CT
* Individuals with bleeding disorders

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1514 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Measuring the positive and negative predictive value of a circulating tumor DNA blood test in detecting the presence of cancer or pre-cancerous lesions | 1-2 years
  Within a year of all blood sample collections, the following will be determined:
  * Number of False Positive Tests - The number of participants with a confirmed positive blood test who participated in a diagnostic evaluation during which no cancer was found.
  * Number of True Positive Tests - The number of participants with a confirmed blood test who participated in a diagnostic evaluation during which a cancer was found.

SECONDARY OUTCOMES:
The enrollment rates for this study | 1-2 years
  Based on the recruitment data from the participants of the BC Generations Project, the participant enrollment rates will be determine quarterly, semi-annually and yearly.
The number of repeated versus sporadic positive test results within a year of the last blood draw. | 1-2 years
  After the last blood draw, data will be analyzed to determine the number of repeated versus sporadic positive test results (i.e. how often does the test provide the same results on separate blood draws from the same individual, versus different results).
The rate of participation in the medical imaging component of the study once a positive test result has been confirmed. | 1-2 years
  After the last blood draw, data will be analyzed to determine the rate of participation in the medical imaging component of the study once a positive test result has been confirmed within a year.
The number of medical imaging scans required per thousand individuals enrolled in the study. | 1-2 years
  After the last blood draw, data will be analyzed to determine how often medical imaging scans were required per thousand of enrolled participants.
The number of participants with abnormal medical imaging scans and of those cohorts, what fraction is cancer found. | 1-2 years
  After the last blood draw, data will be analyzed to determine:
  Of the participants with abnormal medical imaging scans
  * what fraction is conclusively diagnosed with cancer within 2 months.
  * The number of curable cancers found
  * The number of incurable metastatic cancers found
  * The number of participants in whom cancer is found by one year after the blood sample, by any means.

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Nichol, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency- Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Only participants have the option of receiving their own personal data.

REFERENCES:
- [Background] Forbes SA, Bindal N, Bamford S, Cole C, Kok CY, Beare D, Jia M, Shepherd R, Leung K, Menzies A, Teague JW, Campbell PJ, Stratton MR, Futreal PA. COSMIC: mining complete cancer genomes in the Catalogue of Somatic Mutations in Cancer. Nucleic Acids Res. 2011 Jan;39(Database issue):D945-50. doi: 10.1093/nar/gkq929. Epub 2010 Oct 15. PMID 20952405
- [Background] Cancer Genome Atlas Research Network; Weinstein JN, Collisson EA, Mills GB, Shaw KR, Ozenberger BA, Ellrott K, Shmulevich I, Sander C, Stuart JM. The Cancer Genome Atlas Pan-Cancer analysis project. Nat Genet. 2013 Oct;45(10):1113-20. doi: 10.1038/ng.2764. PMID 24071849
- [Background] Punnoose EA, Atwal S, Liu W, Raja R, Fine BM, Hughes BG, Hicks RJ, Hampton GM, Amler LC, Pirzkall A, Lackner MR. Evaluation of circulating tumor cells and circulating tumor DNA in non-small cell lung cancer: association with clinical endpoints in a phase II clinical trial of pertuzumab and erlotinib. Clin Cancer Res. 2012 Apr 15;18(8):2391-401. doi: 10.1158/1078-0432.CCR-11-3148. Epub 2012 Apr 5. PMID 22492982
- [Background] Spindler KL, Pallisgaard N, Vogelius I, Jakobsen A. Quantitative cell-free DNA, KRAS, and BRAF mutations in plasma from patients with metastatic colorectal cancer during treatment with cetuximab and irinotecan. Clin Cancer Res. 2012 Feb 15;18(4):1177-85. doi: 10.1158/1078-0432.CCR-11-0564. Epub 2012 Jan 6. PMID 22228631
- [Background] Misale S, Yaeger R, Hobor S, Scala E, Janakiraman M, Liska D, Valtorta E, Schiavo R, Buscarino M, Siravegna G, Bencardino K, Cercek A, Chen CT, Veronese S, Zanon C, Sartore-Bianchi A, Gambacorta M, Gallicchio M, Vakiani E, Boscaro V, Medico E, Weiser M, Siena S, Di Nicolantonio F, Solit D, Bardelli A. Emergence of KRAS mutations and acquired resistance to anti-EGFR therapy in colorectal cancer. Nature. 2012 Jun 28;486(7404):532-6. doi: 10.1038/nature11156. PMID 22722830
- [Background] Kidess E, Heirich K, Wiggin M, Vysotskaia V, Visser BC, Marziali A, Wiedenmann B, Norton JA, Lee M, Jeffrey SS, Poultsides GA. Mutation profiling of tumor DNA from plasma and tumor tissue of colorectal cancer patients with a novel, high-sensitivity multiplexed mutation detection platform. Oncotarget. 2015 Feb 10;6(4):2549-61. doi: 10.18632/oncotarget.3041. PMID 25575824
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385